CLINICAL TRIAL: NCT03572829
Title: A Prospective, Open-label, Single-arm Study for Efficacy and Safety of Three-drug Antiemetic Regimen to Prevent the Emesis During Radiotherapy With Concurrent Chemoradiotherapy in Locally Advanced HNSCC
Brief Title: Aprepitant for Nause and Vomiting Induced by Chemoradiotherapy in HNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jun-Lin Yi, MD, Vice director of department of radiation oncology, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-RCS-004
Record Dates: First submitted 2018-06-07; First posted 2018-06-28 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Vomiting; Nausea Post Chemotherapy; Head Neck Cancer
MeSH Terms: conditions — Vomiting; Head and Neck Neoplasms | interventions — Aprepitant; Dexamethasone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aprepitant (Experimental): Aprepitant combined with ondansetron and dexamethasone
  Interventions: Drug: Aprepitant

INTERVENTIONS:
Drug: Aprepitant — Intensity-modulated radiotherapy was given to the patients with regimen of 69.96 Gy-73.92 Gy to the gross target volume of nasopharynx,69.96 Gy to the gross target volume of positive nodes, 60.06 Gy the high risk clinical target volume, 50.96 Gy to the low risk clinical target volume. Concurrent chemotherapy is administrated with cisplatin 100mg/m2 at d1, d22, d43 during radiotherapy. Patients receive concurrent aprepitant 125mg, dexamethasone 12mg, and ondansetron 8mg p.o. on day1. AND then patients received aprepitant 80mg, dexamethasone 8mg on day 2-5 at every chemotherapy cycle.
  Other Names: Dexamethasone; Ondansetron

SUMMARY:
To evaluate the safety and efficacy of aprepitant combined with ondansetron and dexamethasone to prevent nausea and vomiting induced by Intensity-modulated Radiotherapy (IMRT) cisplatin-chemotherapy regimen in locally advanced squamous cell carcinoma of head and neck

DETAILED DESCRIPTION:
To evaluate the complete response rate, nause-free rate, vomiting-free rate, and the quality of life of aprepitant combined with ondansetron and dexamethasone for the nausea and vomiting induced by chemoradiotherapy in HNSCC.

ELIGIBILITY:
Inclusion Criteria:

Pathology confirmed squamous cell carcinoma. The primary sites included nasopharynx, mouth, oropharynx, hypopharynx, larynx, nasal cavity and paranasal sinuses; Aged 18 to 70 years old; Stage III-IVB diseases; Eastern Cooperative Oncology Group Performance Status 0-1; Normally functioning of liver, kidney, bone marrow; Concurrent chemoradiotherapy is recommended after multi-disciplinary team discussion; Must be able to swallow tablets; At least 12 weeks lifetime was expected; Fertile male or female patients volunteered to use effective contraception within 90 days of the study period and at the end of study.

Exclusion Criteria:

Nausea and vomiting occurred 24 hours before the start of the chemotherapy; Corticosteroid or benzodiazepines used; Combination Medicine which metabolism through drug-metabolizing enzyme CPY3A4 and CYP2D6; Serious cardiovascular, pulmonary, diabetes, mental and other diseases; Perinatal women or refused to take contraception during treatment; Other induced vomiting factors. (The transfer of the central nervous system, intestinal obstruction or hypocalcemia, and so on)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Complete response rate | up to 8 weeks
  no vomiting and nausea, and no use of rescue therapy

SECONDARY OUTCOMES:
Complete response rate | up to 3 weeks
  no vomiting and nausea, and no use of rescue therapy
Complete response rate | up to 6 weeks
  no vomiting and nausea, and no use of rescue therapy
European Organization for Research on Treatment of Cancer Quality of life questionnaire | up to 12 weeks
  Quality of life questionnaire core 30 chinese version is used. The total score is reported, and the high values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Junlin Yi, M.D., Principal Investigator — National Cancer Center/ Cancer Hospital, Chinese Academy of Medcal science and Peking Union Medical College
Locations (1):
- National Cancer Center/ Cancer Hospital, Chinese Academy of Medcal science and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No